CLINICAL TRIAL: NCT05994911
Title: The Effect of Mindfulness Education on Interpersonal Style and Perceived Social Competence in Adolescents
Brief Title: Mindfulness Education in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ejdane Coskun (Other)
Responsible Party: Sponsor-Investigator, Ejdane Coskun, PhD, Lecturer, Osmaniye Korkut Ata University
Organization: Osmaniye Korkut Ata University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Mindfulness
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Mindfulness
Keywords: Mindfulness Training; Adolescent; Interpersonal Style; Perceived Social Competence; Psychiatric nursing
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Training adolescent (Experimental): An 8-week interview will be conducted with the individuals in the experimental group in the research in which the mindfulness training psychiatric nursing approach is applied. The control group will continue their routine school life. Individuals in the experimental group will be trained as a group and initiatives will be implemented in line with the goals of the individuals and the objectives of the research.
  Interventions: Behavioral: Mindfulness Training
- Mindfulness (No Intervention): Individuals in the control group will continue their school life.

INTERVENTIONS:
Behavioral: Mindfulness Training — The application is planned as 8 sessions and one session per week. Each session corresponds to one lesson hour and is approximately 30-40 minutes. In the content of the application, the individual's attention, mind, attitude, intention, thought; It has basic concepts such as the separation and merging process of thoughts in our minds, the deep processes of awareness, staying in the moment, values, focusing process, self-compassion, integration of awareness with other situations in life, meditation practices developed with practice, and the content summarized around these concepts. It is a program that tries to enable individuals to focus on the moment they live in, within the framework of these basic concepts. The program is divided into session titles such as "Introduction to Mindfulness", "Mind Awareness", "Body Awareness", "Emotion and Behavior Awareness", "Self Compassion", "Stress Awareness", "Eating Awareness".
  Other Names: Mindfulness
  Arms: Mindfulness Training adolescent

SUMMARY:
Aim: It was planned to evaluate the impact of mindfulness training on interpersonal style and perceived social competence in adolescents.

DETAILED DESCRIPTION:
In the research, high school students will form the universe according to the education in the relevant institution. Based on a study with a similar design, it was decided to include 60 people, 30 in the intervention group and 30 in the control group, according to the effect size.

ELIGIBILITY:
Inclusion Criteria:

be a high school student

Exclusion Criteria:

Having any psychiatric illness that prevents adequate communication will not be included in the study.

Ages: 17 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Mindfulness training affects interpersonal style in adolescents. | up to 8 weeks
  It was developed to determine what style they use in interpersonal relationships. It is a self-assessment scale consisting of sixty items. The items are answered according to the question "How much does it describe you" and are answered in a 5-point Likert type as 0%, 25%, 50%, 75% and 100%. 0.1%, 1 point; 25%, 2 points; 50%, 3 points; 75% are evaluated with 4 points and 100% with 5 points. Accordingly, a minimum of 60 and a maximum of 300 points can be obtained.

SECONDARY OUTCOMES:
Mindfulness training affects perceived social competence in adolescents | up to 8 weeks
  The Perceived Social Competence Scale is a one-dimensional scale consisting of 6 items and items. The highest score that can be obtained from the scale is 30, and the lowest score is 6. It can be said that as the scores obtained from the Perceived Social Competence Scale, which does not have any reversed items, increase, the perceived social competency level of the individual also increases

CONTACTS AND LOCATIONS:
Overall Officials: Ejdane Coşkun, Lect., Principal Investigator — Korkut Ata University Osmaniye, Center, Türkiye, 80000; Ayşe İNEL MANAV, Assoc. Prof, Principal Investigator — Korkut Ata University Osmaniye, Center, Türkiye, 80000; Hüsne Demirel, Assoc. Prof, Principal Investigator — Gazi University Ankara, Center, Türkiye, 06500; Yunus Ömer Arık, Grad. stud., Principal Investigator — Korkut Ata University Osmaniye, Center, Türkiye, 80000
Locations (1):
- Türkiye, Osmaniye, Korkut Ata University, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No